CLINICAL TRIAL: NCT02917525
Title: Bicuspid Aortic Valve Stenosis and the Effect of vItamin K2 on Calciummetabolism on 18F-NaF PET/MRI (BASIK2): a Pilot Study
Brief Title: Bicuspid Aortic Valve Stenosis and the Effect of vItamin K2 on Calciummetabolism on 18F-NaF PET/MRI
Acronym: BASIK2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC152045
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Aortic Valve Stenosis; Bicuspid Aortic Valve
Keywords: Calcium metabolism; Matrix Gla Protein; Vitamin K2
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin K2 (Experimental): 22 patients will receive 360ug Vitamin K2 daily during 18 months.
  Interventions: Dietary Supplement: Vitamin K2
- Placebo (Placebo Comparator): 22 patients will receive placebo during 18 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2
  Arms: Vitamin K2
Other: Placebo
  Arms: Placebo

SUMMARY:
Early development of calcified aortic valve disease (CAVD) is a commonly occurring complication in patients with a bicuspid aortic valve (BAV, an aortic valve consisting of two leaflets instead of three). In general, CAVD is characterized by progressive narrowing of the aortic valve, with involvement of altered calcium metabolism. CAVD progression in fact may lead to necessity of valve replacement, since to date, no other therapies have been shown effective in the treatment of CAVD.

The primary objective of our study is to test the hypothesis that supplementation of vitamin K2 will slow down the calcium metabolism in CAVD. Vitamin K2 is essential in the activation of matrix Gla Protein (MGP), an important inhibitory factor in the regulation of calcification.

In this randomized controlled trial, 44 patients will be allocated to either the vitamin K2 or placebo group. To assess the calcification process in a detailed manner in these patients, a Positron Emission Tomography (PET) scanner using a tracer (18F-fluoride [NaF]) that has been shown to bind to regions of newly developing microcalcification in aortic valve tissue is used.

We expect that vitamin K2 supplementation will reduce the calcium metabolism in the aortic valve on 18NaF-PET (primary endpoint) and slow progression of CAVD as measured by the calcium score on CT and echocardiography after 18 months (secondary endpoints), when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* known bicuspid aortic valve
* calcified mild to moderate aortic valve stenosis on prior echocardiography
* informed consent provided

Exclusion Criteria:

* absence of calcified aortic valve stenosis on echocardiography
* presence of severe aortic valve stenosis
* history of aortic valve repair or replacement
* accepted atrial fibrillation
* use of oral anticoagulants
* claustrophobia
* presence of a pacemaker, ICD or ferromagnetic materials in the body
* life expectancy <2 years
* Pregnancy (current or wish for near future)
* soy allergy
* use of vitamin K-containing supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in aortic valve calcium metabolism | Measured at baseline and 6 months
  Change in calcium metabolism, measured as uptake of the 18F-NaF tracer on a 18F-NaF PET/CMR scan

SECONDARY OUTCOMES:
Change in aortic valve calcium score | Measured at baseline, 6 and 18 months
  Change in aortic valve calcium score, measured on CT.
Progression of aortic valve stenosis | Measured at baseline, 6, 12 and 18 months
  Change of severity of aortic valve stenosis on echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Bas Kietselaer, M.D. PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Netherlands